CLINICAL TRIAL: NCT05651568
Title: Comparison of Periodized Resistance Training and High Intensity Interval Training on Body Mass Index and Quality of in Polycystic Ovarian Syndrome.
Brief Title: Effect of Periodized Resistance Training and High Intensity Training on BMI and QOL in PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Adeela Arif
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodized resistance training (Experimental): It consists of patients who will receive periodized resistance training 3 sessions per week for 8 weeks. Resistance training has been performed according to FITT principal and as per ACSM recommendation.
  Interventions: Other: Periodized resistance training
- High intensity interval training (Experimental): It consists of patients who will receive high intensity interval training 3 sessions per week for 8 weeks for 30-35 minutes.
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: Periodized resistance training — It consists of patients who will receive periodized resistance training 3 sessions per week for 8 weeks. Resistance training has been performed according to FITT principal and as per ACSM recommendation.
  Frequency:
  Three days in a week
  Intensity:
  60% intensity with one repetition maximum and 10% intensity were added each the two weeks.4 sets and 8-12 rep as per ACSM criteria. There will be rest of 60 second after every set and 120 seconds after every exercise.
  Type:
  8 types of resistance exercises were performed. There were 4 set of each exercise with 8 to 12 repetitions. These exercises are smith press, seated press, squat, lying dumbbell leg curls, leg extension, leg press, standing barbell, lying barbell and sit ups.
  Time:
  40 minutes per session.
  Arms: Periodized resistance training
Other: High intensity interval training — It consists of patients who will receive high intensity interval training 3 sessions per week for 8 weeks for 30 to 35 minutes.
  Active phase: Two weekly sessions of four times four minutes at 90-95% of individual heart rate maximum, separated by three minutes of active rest period and one weekly session of ten times one minute with maximal intensity, separated by one minute of active rest. The exercise mode will be treadmill or outdoor walking/running or cycling (self-selected).
  Arms: High intensity interval training

SUMMARY:
This study may help to improve strength and body composition in females with PCOS. It will enhance ability of an overweight individual to perform functional tasks (i.e. daily living tasks or physical activity) to be physically active. This may facilitate the adoption of a more active lifestyle, thereby increasing the likelihood of success in overall weight-reduction strategies.

DETAILED DESCRIPTION:
Poly cystic ovarian syndrome (PCOS) is a hormonal disorder which is most common in females with fertile age. A number of small fluid filled sacs formed in ovaries which results in failure of egg release. Poly cystic ovary syndrome (PCOS) is an endocrine problem which is characterized by the polycystic ovaries, menstrual problems, infertility, metabolic disorder, psychological problems, elevated androgens, hirsutism, acne and obesity. PCOS also causes psychological disorders which include depression, anxiety, poor body image, low self-esteem and decreased health- related quality of life. Some well-controlled randomized clinical studies have been conducted to evaluate the effects of exercise training program in women with PCOS. There are many beneficial effects of exercises which improve physical fitness, body composition, and cardiovascular, hormonal, reproductive and psychological outcomes. Periodization training program involves period of active rest which allows muscle adaptations through variable intensity, volume and rest. The advantage of periodization is that it prevent from overtraining symptoms such as muscle stiffness, muscle soreness, sprain, strain, possible injury and decreased performance. High intensity interval training is effective in reducing body mass index and improving body composition in females with PCOS.

The study will be a randomized clinical trial and will be conducted in Mohsin memorial hospital Faisalabad. This study will be completed in time duration of ten months after the approval of synopsis and convenient sampling technique will be used. Total twenty four subjects will be assigned randomly by using lottery method into two groups. Group A will receive periodized resistance training and Group B will receive high intensity interval training. Warm up and cool down period of ten minutes of treadmill training will be performed by both groups. Data will be collected from all participants at baseline and after 8 weeks of treatment by using BMI and WHO-QOL BREF questionnaire. After assessing the normality data will be analyzed by using parametric or non-parametric test by using SPSS-25.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-35 years
* Unmarried females
* Diagnosed patients of PCOS
* All women who are less physically active or have sedentary life style.
* BMI>25kg/m2 (overweight obese)

Exclusion Criteria:

* Use of hormonal contraceptives.
* Diabetes
* Hypertension
* Thyroid disease
* Cushing disease
* Any physical disability

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 8th week
  Body mass index is a screening tool derived from the weight and height of a person. It is a simple numeric measure of a subject"s thickness or thinness. Calculated values help in determining if a person is underweight, normal weight or overweight. Body mass index used to classify average sedentary (physically inactive) populations, with an average body composition. Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in meters squared. A BMI of 25.0 or more is overweight, while the healthy range is 18.5 to 24.9.
WHO quality of life Bref | 8th week
  The WHOQOL- BREF is a 26 items self-report questionnaire consisting of 4 domains of quality of life. Physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains 2 items of overall QOL and general health.

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Arif, Mphil, Principal Investigator — Riphah International University
Locations (1):
- PSRD, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christodoulopoulou V, Trakakis E, Pergialiotis V, Peppa M, Chrelias C, Kassanos D, Papantoniou N. Clinical and Biochemical Characteristics in PCOS Women With Menstrual Abnormalities. J Family Reprod Health. 2016 Dec;10(4):184-190. PMID 28546817
- [Background] Venkatesh SS, Ferreira T, Benonisdottir S, Rahmioglu N, Becker CM, Granne I, Zondervan KT, Holmes MV, Lindgren CM, Wittemans LBL. Obesity and risk of female reproductive conditions: A Mendelian randomisation study. PLoS Med. 2022 Feb 1;19(2):e1003679. doi: 10.1371/journal.pmed.1003679. eCollection 2022 Feb. Erratum In: PLoS Med. 2022 Sep 2;19(9):e1004095. doi: 10.1371/journal.pmed.1004095. PMID 35104295
- [Background] Jobanputra H, Pawar V, Guhe A, Kalambe SRNM, Chaudhary A. Polycystic Ovarian Syndrome with Physical Therapy Management and A Proof-Primarily Based Totally Evaluation Article for Exercise in Pcos. NVEO-NATURAL VOLATILES & ESSENTIAL OILS Journal| NVEO. 2021:1370-81.
- [Background] Clemente-Suarez VJ, Ramos-Campo DJ. Effectiveness of Reverse vs. Traditional Linear Training Periodization in Triathlon. Int J Environ Res Public Health. 2019 Aug 6;16(15):2807. doi: 10.3390/ijerph16152807. PMID 31390818